CLINICAL TRIAL: NCT03611400
Title: The Effect of Probiotic Intake on Intestinal Permeability of Healthy Adults
Brief Title: The Effect of Probiotic Intake on Intestinal Permeability in Healthy Adults
Acronym: PIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: IRB201800616; OCR18441 (Other: University of Florida)
Record Dates: First submitted 2018-06-27; First posted 2018-08-02 (Actual); Last update posted 2019-06-21 (Actual); Status verified 2019-06

CONDITIONS: Intestinal Barrier Function
Keywords: Probiotic; Intestinal Permeability; Leaky Gut
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Intervention Model Description: A randomized, double-blind, placebo-controlled crossover in which participants receive one of the study supplements (probiotic or placebo) for a 3-week intervention period each will be used.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participants, investigators, and anyone else involved with the study will remain blinded for its entirety.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotic (Experimental): 2 capsules daily for 3 weeks, containing 3.8 x 10^9 CFU (colony forming units)/capsule of Lactobacillus rhamnosus strain R011and 0.2 x 10^9 CFU/capsule of L. helveticus strain R0052 (group is unknown, double blinded)
  Interventions: Dietary Supplement: Probiotic
- Placebo (Placebo Comparator): 2 capsules daily for 3 weeks containing the same carrier material and is similar in size, shape and taste to probiotic (group is unknown, double blinded)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic — This probiotic is commercially available and contains L. helveticus R0052 (0.2 x 10^9 CFU/capsule) and L. rhamnosus R0011 (3.8 x 10^9 CFU/capsule) as active ingredients and ascorbic acid, hypromellose, magnesium stearate, saccharose, potato starch, titanium dioxide, and maltodextrin as excipients.
  Other Names: Lacidofil STRONG
  Arms: Probiotic
Dietary Supplement: Placebo — The placebo contains ascorbic acid, hypromellose, magnesium stearate, saccharose, potato starch, titanium dioxide and maltodextrin.
  Arms: Placebo

SUMMARY:
In this double blind, crossover study participants will take a placebo for 3 weeks each. Gut permeability will be assessed weekly using food-grade sugar molecules. On the second week, participants will take aspirin, which will make their intestine permeable to the sugars. Participants will be asked to provide urine and stool samples to assess gut permeability and microbial communities. No change in permeability to the small sugar probes is anticipated with the probiotic.

ELIGIBILITY:
Inclusion Criteria

1. Healthy individuals, aged 21 to 50 years who have ≥6 stools/week.
2. Willing to discontinue the use of non-steroidal anti-inflammatory drugs (NSAIDs), such as ibuprofen, aspirin, naproxen, or indomethacin, for the full length of the study.
3. Willing to avoid beer, wine, and cocktails on the day before and the day of the sugar probe tests. The sugar probe tests are visits 2, 3, 4, 6, 7, and 8.
4. Willing to avoid the use of antidiarrheal or laxative medication on a regular or an "as-needed basis" during the full length of the study.
5. Willing to provide urine and stool samples during the study collection periods.
6. Have used aspirin in the past and did not experience adverse effects.
7. Willing to consume three tablets (325 mg each or 975 mg total) twice within a 9 to 12-hour period. This challenge will be repeated twice during the 14-week study.
8. Willing to complete online questionnaires, records, and diaries associated with the study and to complete all clinic visits.
9. Willing to discontinue consumption of fermented foods or probiotics.
10. Willing to discontinue taking prebiotic, herbal, or high-dose vitamin or mineral supplements that may impact immune function or inflammation during the pre-baseline period and throughout the study protocol.
11. Willing to avoid high intensity exercises two days prior to and the day of the permeability tests. These tests will be done on six occasions.
12. Willing and able to consume the probiotic and placebo daily for 3 weeks each.
13. Willing and able to complete the informed consent form in English.
14. Willing to provide a social security number to receive study payment.

Exclusion Criteria

1. History or current impaired cardiovascular circulation or uncontrolled hypertension, diabetes, bleeding tendencies, kidney, liver or chronic respiratory diseases including asthma, gastrointestinal disorders including heartburn, or any other disease, that by the investigators discretion could interfere with the intestinal barrier function of the subject.
2. Daily use of NSAIDs in the last 3 months or incidental use in the last 2 weeks prior to screening.
3. Use of medications in the last 2 weeks prior to the pre-baseline period. This does not include birth control pills or standard multi-vitamin/mineral supplements.
4. Allergy to aspirin, milk, yeast, or soy.
5. Known sensitivity to gluten.
6. Current smokers.
7. Women who are lactating, know that they are pregnant, or are attempting to get pregnant.
8. Use of another investigational product within 3 months of the screening visit.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2018-08-22 (Actual); Primary Completion 2019-04-15 (Actual); Study Completion 2019-04-15 (Actual)

PRIMARY OUTCOMES:
Gastroduodenal Permeability | Week 2 of each intervention
  The primary outcome is the difference between the changes in gastroduodenal permeability induced by aspirin challenge with the probiotic versus the placebo. Gastroduodenal permeability will be assessed while on the placebo and probiotic interventions by measuring urinary sucrose in the 0 to 5-hour urine collection of the sugar probe permeability test. Change will be calculated as the urinary sucrose concentration after aspirin challenge (week 2 of each intervention) minus the concentration from the prior week (i.e., 1 wk on intervention with no aspirin challenge).

SECONDARY OUTCOMES:
Small Intestinal Permeability | Weeks 1 and 2 on intervention
  Difference between the changes (week 2 of intervention with aspirin minus week 1 of intervention without aspirin) in urinary lactulose/rhamnose ratio in the 0 to 5-hour urine collection with the probiotic versus the placebo interventions.
Colonic Permeability | Weeks 1 and 2 on intervention
  Difference between the changes (week 2 of intervention with aspirin minus week 1 of intervention without aspirin) in sucralose/erythritol ratio in the 5 to 24-hour urine collection with the probiotic versus the placebo interventions.
Whole Gut Permeability | Weeks 1 and 2 on each intervention
  difference in the changes (week 2 of intervention with aspirin minus week 1 of intervention without aspirin) in sucralose/erythritol ratio in the 0 to 24-hour urine collection with the probiotic versus the placebo interventions

OTHER OUTCOMES:
Digestive Health | Weekly through the completion of the 14 week study
  Weekly GI symptoms assessed using the Gastrointestinal Symptom Rating Scale (GSRS). The GSRS consists of 15 questions related to 5 syndromes, constipation, diarrhea, reflux, abdominal pain, and indigestion. Symptoms are scored 1=no discomfort to 7=very severe discomfort. Scores from each of the 15 questions are summed for the total GSRS score.

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No